CLINICAL TRIAL: NCT06144320
Title: The Objective of Our Study is to Evaluate the Medium and Long-term Clinical Efficacy of Acupuncture in Patients With Post Covid Related Mild Cognitive Impairment (MCI).
Brief Title: Efficacy of Acupuncture in Patients Post-Covid Brain Fog
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chien Yu Huang, doctor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH112-REC2-108
Record Dates: First submitted 2023-11-21; First posted 2023-11-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-07

CONDITIONS: Brain Fog
Keywords: Brain fog
MeSH Terms: conditions — Mental Fatigue | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Practicing acupuncture on specific acupoints. The retention time of the needle is 30 minutes every time and the frequency of treatment is 3 times per week for 8 weeks.
  Interventions: Other: Acupuncture
- Placebo group (Sham Comparator): Practicing sham acupuncture on specific acupoints is the same as the treatment group, and also the same retention and frequency.
  This study used the specifically made needle with a blunt tip, the Streitberger device, as the sham acupuncture. The needle does not penetrate the skin and retracts in the handle while the acupuncturist needles into the skin.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture is performed using acupuncture points recorded in traditional Chinese medicine books as helpful for cognitive impairment.

SUMMARY:
After being infected with Covid-19, many people developed to Brain fog. The treatment strategy now is based on the presumed pathological phenomenon and the physician's clinical experience. Acupuncture has been used to improve cognitive dysfunction caused by central nervous system diseases for many years.

A randomized rater-blinded controlled study is proposed to see the efficacy of acupuncture for brain fog.

DETAILED DESCRIPTION:
After being infected with Covid-19, many people develop cognitive dysfunction, including deficits in attention, executive ability, language, processing speed, and memory. These symptoms are collectively known as Brain fog or Covid fog.

The pathological mechanism of the cognitive deficit is inconclusive. Therefore, the treatment strategy is based on the presumed pathological phenomenon and the physician's clinical experience. Acupuncture has been used to improve cognitive dysfunction caused by central nervous system diseases for many years. This study aims to evaluate the medium and long-term clinical efficacy of acupuncture in patients with post-Covid related Mild cognitive impairment (MCI).

A randomized rater-blinded controlled study is proposed. Eligible patients were over 18 years old and <65 years old. These patients were diagnosed with Covid-19 more than 12 weeks earlier and developed mild cognitive impairment (MCI) after the diagnosis of Covid-19. Divided into the acupuncture group and the sham acupuncture group for an 8-week course of treatment, the Mini-Mental State Examination (MMSE), the quality of life assessment scale The 5-level EQ(EuroQol Group)- five dimensions version(EQ-5D-5L) and The Stroop Color and Word Test evaluates the degree of cognitive impairment and the impact of cognitive impairment on quality of life and attention.

ELIGIBILITY:
Inclusion Criteria:

1. Have been tested positive for severe acute respiratory syndrome coronavirus 2(SARS-CoV-2) or had serum antibody positivity more than 12 weeks before.
2. Present cognitive impairment after been diagnosed as Covid-19
3. Clinical Dementia Rating (CDR) score of 1
4. Normal activities of daily living score (ADL)
5. (Mini-Mental State Examination) MMSE score of 24-28
6. Age of 18-65 years
7. Signed informed consent

Exclusion Criteria:

1. Diagnosed with any type of dementia.
2. A history of acute or chronic cerebrovascular disease, encephalitis, Parkinson's disease, Leukoencephalopathy, and other central nervous system diseases
3. A history of hypothyroidism, vitamin B12 deficiency, depression, syphilis, and other diseases that may affect cognitive decline.
4. Severe hearing and visual impairment, inability to complete neuropsychological tests
5. Impaired liver and kidney function and hematopoietic system disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
cognitive function | The measurement is assessed before the first treatment, and recheck on 4th,8th week and 4 weeks after finishing the course of treatment.
  Mini-Mental State Examination (MMSE) is used to assess include orientation, memory, calculation ability and attention, information registration, operational ability, language comprehension, spatial concepts.

SECONDARY OUTCOMES:
Concentration difficulty | The measurement is assessed before the first treatment, and recheck on 4th,8th week and 4 weeks after finishing the course of treatment.
  The Stroop Color and Word Test (SCWT) was chosen to evaluate the changes in attention.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leng A, Shah M, Ahmad SA, Premraj L, Wildi K, Li Bassi G, Pardo CA, Choi A, Cho SM. Pathogenesis Underlying Neurological Manifestations of Long COVID Syndrome and Potential Therapeutics. Cells. 2023 Mar 6;12(5):816. doi: 10.3390/cells12050816. PMID 36899952
- [Result] Seessle J, Waterboer T, Hippchen T, Simon J, Kirchner M, Lim A, Muller B, Merle U. Persistent Symptoms in Adult Patients 1 Year After Coronavirus Disease 2019 (COVID-19): A Prospective Cohort Study. Clin Infect Dis. 2022 Apr 9;74(7):1191-1198. doi: 10.1093/cid/ciab611. PMID 34223884
- [Result] Venkataramani V, Winkler F. Cognitive Deficits in Long Covid-19. N Engl J Med. 2022 Nov 10;387(19):1813-1815. doi: 10.1056/NEJMcibr2210069. No abstract available. PMID 36351274
- [Result] Kao J, Frankland PW. COVID fog demystified. Cell. 2022 Jul 7;185(14):2391-2393. doi: 10.1016/j.cell.2022.06.020. Epub 2022 Jun 15. PMID 35768007
- [Result] Lempriere S. Inflammation links mild COVID-19 with long-term cognitive impairment. Nat Rev Neurol. 2022 Aug;18(8):453. doi: 10.1038/s41582-022-00694-x. PMID 35773475